CLINICAL TRIAL: NCT01883791
Title: Screening, Brief Intervention and Referral to Treatment for Substance Abuse in Mental Health Treatment Settings
Acronym: SBIRT in MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Suzette Glasner-Edwards, Research Psychologist, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01DA032733-01A1 (NIH); R01DA032733 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2013-06-21 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Substance Use Disorders; Mental Illness
Keywords: substance abuse prevention and treatment; comorbidity; SBIRT
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders | interventions — Mass Screening; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBIRT (Experimental): The SBIRT condition will include the WHO's Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) and its accompanying brief intervention that uses motivational interviewing techniques to provide feedback, emphasize personal responsibility, give advice, provide a menu of options, convey empathy, and promote self-efficacy.
  Interventions: Behavioral: SBIRT
- Health Education (Other): The control group will receive a Health Education (HE) session, informational brochures and a contact information for addiction treatment sites that we will develop with Ventura County. The session will be administered in an individual format for 30-minutes and will address general health, wellness and lifestyle topics.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: SBIRT — See above Arm description.
  Other Names: Screening, Brief Intervention and Referral to Treatment.
  Arms: SBIRT
Behavioral: Health Education — See Arm Description.
  Arms: Health Education

SUMMARY:
An estimated 40% of patients in mental health treatment settings engage in hazardous alcohol and/or drug use. One model of intervention that has been shown effective in medical settings to reduce alcohol use and/or promote engagement in addiction treatment is screening, brief intervention, and referral to treatment (SBIRT). Despite the effectiveness of SBIRT for risky alcohol use in medical settings, there has been no research on the effectiveness of SBIRT in mental health treatment settings. Given the proportionately large number of mental health patients who also engage in hazardous substance use, research is needed to find an appropriate and effective substance use intervention for patients in these settings.

The proposed study uses a randomized controlled trial to examine the extent to which the World Health Organization's SBIRT model, the ASSIST (Alcohol, Smoking, and Substance Involvement Screening Test) and its associated brief behavioral intervention, leads to reductions in substances prevalent in mental health settings: alcohol, cannabis and stimulants (i.e., cocaine and methamphetamine). The study will also examine the effect of SBIRT on improvement in psychiatric symptoms, improved quality of life and for those whose level of substance misuse indicates a need for treatment, initiation and engagement into SUD treatment services. Eligible participants will be mental health patients who report any past year use of cannabis or stimulants or at least one heavy drinking day in the past year. Mental health patients (N=750) who meet eligibility criteria will be enrolled and randomly assigned to either the SBIRT intervention condition or to a health education attention control condition. Participants will be assessed at baseline on substance use, psychiatric symptoms and quality of life. Each participant will be assessed at 3-, 6- and 12- month follow up points for alcohol and drug use, involvement in SUD treatment services, severity of psychiatric symptoms and quality of life. If successful this study will yield valuable new knowledge about the effectiveness of SBIRT in mental health treatment settings and will promote improved well being of mental health patients. Further, the study will provide evidence on the effectiveness of SBIRT for reducing illicit drug use. Results from this research will be used as the basis for broader dissemination and of SBIRT in mental health settings.

DETAILED DESCRIPTION:
Research Design and Methods The proposed 5-year study is a randomized, controlled trial of screening, brief intervention, and referral to treatment (SBIRT) for alcohol, cannabis and stimulant use in mental health treatment settings. These 3 substances have been chosen as the focus for the proposed study because (a) in the US alcohol and cannabis are the most common substances used by individuals with serious mental illness in the general population1 and (b) stimulant use (in particular, methamphetamine) is a significant public health threat in the US. 31,32 The SBIRT model will be tested in a two-group design in which eligible participants (N=750) will be randomly assigned to either the SBIRT intervention condition (N=375) or to a control condition (N=375) that offers an informational leaflet. The participants will comprise male and female mental health patients who have a positive pre-screen for being at risk of having or developing a substance use disorder. The performance site for the study will be publicly-funded mental health clinics in Ventura County, California. All participants (intervention and control groups) will receive mental health care as usual and their participation in the study will in no way reduce the level of usual care they receive.

The SBIRT condition will include the WHO's Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) and its accompanying brief intervention that uses motivational interviewing techniques to provide feedback, emphasize personal responsibility, give advice, provide a menu of options, convey empathy, and promote self-efficacy.33,34 All participants in the SBIRT condition will complete the ASSIST as an interview. Based on the results of the ASSIST, participants who score in the moderate-risk range for alcohol, cannabis or a stimulant will immediately receive a 15-minute brief intervention. Participants who score in the high-risk range for one of these substances will receive the brief intervention and a referral to a substance abuse treatment facility for further assessment and rehabilitative care. Referral to treatment will be an active intervention and is described below in 'Description of Study Conditions'. We expect that few patients will score in the low-risk range on the ASSIST because the pre-screen for the study (described below in 'Recruitment of Participants and Randomization') should exclude most of these individuals. In the event that any individuals enroll in the study and score in the low-risk range on the ASSIST, their data will be excluded from analysis and they will not be counted toward the target enrollment for the study.

The baseline assessment will occur prior to randomization. Research assistants will administer the assessments in-person at each clinic. Clinical social workers (English and Spanish speaking) will conduct the SBIRT intervention with patients. Follow-up assessments will occur at 3-, 6- and 12-months post baseline.

Project Timeline Table 1 summarizes the main study activities across the 5 years of the project. The research and clinical facilities are in place, but a start-up period of 6 months will be needed to complete the IRB application and approval process, develop data collection templates, train staff and finalize the study protocols and procedures. As shown below in Table 1, subject recruitment will begin in month 7 and extend for 36 months. The timetable for the project is based on an enrollment of 30 participants per month. This rate of recruitment is feasible based on consultations with the mental health treatment sites and will allow for recruitment of 750 participants into the study. As Table 1 shows, the timeline provides adequate time to collect 12-month follow-up data and conduct data analysis.

Table 1: Project Timeline Months 1-6: Training & start-up activities Months 7-42: Recruitment, SBIRT intervention, & follow-up activities. 30 Participants recruited/month (N=1080) Months 43-54: Complete follow-up activities Months 55-60: Data Analysis, Report Writing

ELIGIBILITY:
Inclusion Criteria. Participants who:

* (1)have affective disorder (Major Depressive Disorder, Dysthymia, Bipolar Disorder) or psychotic disorder (Schizophrenia, Schizoaffective, or Psychotic Disorder Not Otherwise Specified),
* (2) have any use of cannabis or stimulants in the past year or a heavy drinking day (5+/4+ drinks for men/women) in the past year,
* (3) are 18 years or older,
* (4) have a stable living situation (i.e., has not been homeless during the past two years),
* (5) are not under the influence of alcohol and/or drugs at the time of enrollment and
* (6) have not received substance abuse treatment within the past year.

Exclusion Criteria. Patients who:

* (1) have received any substance abuse treatment in the past year will be excluded because exposure to addiction treatment may confound the effects of the SBIRT intervention.
* (2) have Opiate and opioid use because we cannot guarantee access to appropriate pharmacotherapies (e.g., suboxone or methadone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back (TLFB) | These data will be assessed for each 90-day period preceding the 3-, 6- and 12-month follow ups.
  The TLFB will be used to determine days of use for alcohol and drugs over the 90-day period prior to the baseline assessment. The interviewer will guide the participant to identify the number of standard drinks consumed each day, starting from the day immediately before the assessment and moving backwards in time. Days on which cannabis and/or stimulants were used will also be queried. Variables calculated from the interview will include: (1) total standard drinks, (2) drinking frequency, (3) heavy-drinking frequency (5+ for men; 4+ for women), (4) maximum quantity of alcohol consumed, (5) number of days using cannabis, (6) number of days using cocaine, (7) number of days using methamphetamine, and (8) days on which any alcohol, cannabis or stimulant was used. This measure is completed at 3, 6 and 12 months post baseline in order to measure change from one timepoint to the next.

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Karno, Ph.D., Principal Investigator — University of California, Los Angeles; Suzette Glasner-Edwards, Ph.D., Principal Investigator — University of California, Los Angeles; Richard Rawson, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Inpatient and Outpatient Psychiatric Units, Los Angeles, California
  - Ventura County Behavioral Health, Oxnard, California